CLINICAL TRIAL: NCT02651935
Title: A Randomized Controlled Trial Comparing a Fully Closed Loop Ventilation Mode (Intellivent ASV) With Pressure Controlled + Pressure Support Ventilation in COPD Patients
Brief Title: Intellivent ASV in Chronic Obstructive Pulmonary Disease Patients in the ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Cenk Kirakli, M.D., Associate Professor, Pulmonary and Critical Care Medicine, Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IGHCEAH-ICU-3
Record Dates: First submitted 2015-02-06; First posted 2016-01-11 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Respiration, Artificial; weaning; critical care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intellivent ASV (Experimental): Patients in this arm will be ventilated with Intellivent ASV. Intellivent ASV is an automatic close loop ventilation mode. FiO2 setting will be automatically adjusted according to patients SpO2 and minute volume will be automatically adjusted according to patients EtCO2.
  Interventions: Device: Intellivent ASV
- PCV+PSV (No Intervention): PCV+PSV is a conventional ventilation strategy of pressure controlled ventilation PCV) and pressure support ventilation (PSV).In this arm, FiO2, pressure control levels, respiratory frequency and all the ventilator settings will be manually adjusted by the physicians in charge.

INTERVENTIONS:
Device: Intellivent ASV — Automated Invasive mechanical ventilation and weaning strategy
  Arms: Intellivent ASV

SUMMARY:
This study will evaluate the effect of a fully closed loop ventilation mode (Intellivent ASV) on the duration of ventilation compared to conventional modes in COPD patients.

DETAILED DESCRIPTION:
COPD patients often need invasive mechanical ventilation and due to the difficulties in the weaning of these patients, duration of mechanical ventilation can be relatively longer when compared with other ICU patients. Automated systems show promising results in shortening the weaning time in some patient groups. The aim of this study is to evaluate the effect of Intellivent-ASV with Quickwean function on the total duration of invasive mechanical ventilation as a primary outcome. Secondary outcomes are success rate and duration of weaning, ventilator free days at day 28 and intubation free days at day 28 (including NIV) when compared to conventional ventilation with t-piece weaning.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients intubated and mechanically ventilated for less than 24 hours (Including patients who received NIV before intubation)
* Age > 18 years
* Written and/or informed consent

Exclusion Criteria:

* Septic shock
* Tracheostomy and/or home mechanical ventilation
* Expected poor short term prognosis
* Cardiac arrest with a poor neurological prognosis
* ARDS
* Broncho-pleural fistula

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-08; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Duration of intubation | 24th month
  Time from intubation until extubation
Duration of mechanical ventilation (NIV included) | 24th month
  Total time patient remains on mechanical ventilation support (invasive or noninvasive)

SECONDARY OUTCOMES:
Number of manual settings | 24th month
  Number of adjusments made manually to set the ventilator
Number of blood gas analysis tests | 24th month
  Number of arterial blood gas tests under mechanical ventilation
Weaning duration | 24th month
  Time from the beginning of weaning until extubation
Time spent on spontaneous ventilation | 24th month
  Time patient actively triggers the ventilator

CONTACTS AND LOCATIONS:
Overall Officials: Ilknur Naz, Principal Investigator — Izmir Chest Diseases and Surgery Training Hospital; Burcu CINLETI, Principal Investigator — Izmir Chest Diseases and Surgery Training Hospital; Huseyin OZKARAKAS, Principal Investigator — Izmir Chest Diseases and Surgery Training Hospital; Tunzala YAVUZ, Principal Investigator — Izmir Chest Diseases and Surgery Training Hospital
Locations (1):
- Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital, Intensive Care Unit, Izmir, Turkey (Türkiye)